CLINICAL TRIAL: NCT06829654
Title: Safety Assessment Of Cryopreserved Ovarian Tissue Transplantation In Patients Who Have Survived Sarcomas And Hematological Tumors
Brief Title: Cryopreserved Ovarian Tissue Transplantation in Patients Who Have Survived Sarcomas and Hematological Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CRIOTESOVA2024
Record Dates: First submitted 2025-01-10; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Sarcomas; Haematological Malignancies
Keywords: sarcomas; haematological malignancies; cryopreservation; ovarian tissue
MeSH Terms: conditions — Sarcoma | interventions — SE 1-step Futurabond M

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients who request cryopreservation of ovarian tissue (Other): Patients who request cryopreservation of ovarian tissue
  Interventions: Other: Step 1; Other: Step 2; Other: Step 3
- Patients with already cryopreserved ovarian tissue at the criobank (Other): Patients with already cryopreserved ovarian tissue at the criobank
  Interventions: Other: Step 2; Other: Step 3
- Patients who request ovarian tissue reimplantation (Other): Patients who request ovarian tissue reimplantation
  Interventions: Other: Step 2; Other: Step 3; Other: Step 4

INTERVENTIONS:
Other: Step 1 — Cryopreservation of ovarian tissue
  Arms: Patients who request cryopreservation of ovarian tissue
Other: Step 2 — Analysis of tumor markers in the primary tumor
Other: Step 3 — Search for neoplastic cells in cryopreserved ovarian tissue
Other: Step 4 — Cryopreserved ovarian tissue autotransplantation
  Arms: Patients who request ovarian tissue reimplantation

SUMMARY:
The study aims to test for the presence or absence of primary tumor-specific tumor markers in ovarian tissue. Therefore, there will be a first phase in which pathology-specific markers will be identified in the patients' diagnostic pathological material by histological, immunohistochemical, and molecular analysis; then, tumor markers will be sought in cryopreserved ovarian tissue.

DETAILED DESCRIPTION:
Standardized strategies for detecting neoplastic cells in ovarian tissue of patients with prior sarcomas or oncohematologic malignancies are not available. To increase the safety of ovarian tissue transplantation, the use of advanced and highly sensitive molecular approaches could greatly improve the detection of malignant cells in ovarian tissue.

The study aims to test for the presence or absence of primary tumor-specific tumor markers in ovarian tissue. Therefore, there will be a first phase in which pathology-specific markers will be identified in the patients' diagnostic pathological material by histological, immunohistochemical, and molecular analysis; then, tumor markers will be sought in cryopreserved ovarian tissue.

Identifying highly sensitive molecular tests would lead to increased safety of transplantation in patients cured of sarcomas and oncohematologic diseases. Overall, applications of the techniques under study would increase the chances of resolving infertility, which often reduces the quality of life of these patients, by offering them the chance to procreate and have biological children. The hope of motherhood is an important psychological support and can greatly help patients cope with the difficult treatment process while minimizing social/psychological support. In the long journey of treatment to defeat the disease, being able to offer an option to at least combat the fear of losing endocrine and reproductive function can have a profound impact not only on the patients themselves, but on the entire family and non-family environment.

ELIGIBILITY:
Inclusion Criteria:

For all groups:

* Patients with Ewing (ES) and synovial (SS) sarcoma, acute lymphoblastic leukemia (LLA), acute myeloid leukemia (LMA), chronic myeloid leukemia (LMC) and myelodysplasia (MDS)
* No objection to the procedure of sampling for cryopreservation or reimplantation of ovarian tissue by the patient's reference oncologist (according to PA105)
* Obtaining informed consent.

Group 1:

* Age >18 and under 38 at the time of cryopreservation
* Request for cryopreservation of ovarian tissue at the Laboratory Cryopreservation Ovarian Tissue and Cell Cultures/Criobank IRCCS AOUBO

Group 2:

* Age >18 years
* Ovarian tissue already collected and cryopreserved at the Laboratory for Cryopreservation of Ovarian Tissue and Cell Cultures/Criobank IRCCS AOUBO

Group 3

* Age > 18 years
* Request for reimplantation of cryopreserved ovarian tissue at the Laboratory for Cryopreservation of Ovarian Tissue and Cell Cultures/Criobank IRCCS AOUBO
* Early menopause or menstrual irregularities

Exclusion Criteria:

Group 1 and 3

* Contraindications to laparoscopy
* HIV, hepatitis B and C, treponema pallidum and positive PAP tests
* Malignant disease involving the ovary or samples to be reimplanted

Group 2 None.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of cancer cells on cryopreserved ovarian tissue | through study completion, an average of 1 year
  Detection rate of cancer cells on cryopreserved ovarian tissue for a diagnostic panel specific to pathology in anamnesis, patients with Ewing sarcoma (SE), synovial sarcoma (SS), acute lymphoblastic leukemia (LLA), acute myeloid leukemia (AML), chronic myeloid leukemia (CML) or myelodysplasia (MDS)

SECONDARY OUTCOMES:
Concordance of histological/molecular investigations | through study completion, an average of 1 year
  Establish the correlation between histological-immunohistochemicals investigations and molecular investigations and between molecular investigations in identifying neoplastic cells in cryopreserved ovarian tissue
Disease-specific detection rate | through study completion, an average of 1 year
  Identify the diagnostic method with the highest detection rate for each pathology analyzed, including histo-immunohistochemical investigations and molecular investigations
Ovarian contamination | through study completion, an average of 1 year
  Estimate, for molecular analysis methods, the proportion of ovarian contamination by cancer cells in different pathologies

CONTACTS AND LOCATIONS:
Overall Officials: Renato Seracchioli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy